CLINICAL TRIAL: NCT05963763
Title: Pathways to Economic Mobility Pilot
Brief Title: Economic Mobility Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a shift in organizational factors this study will not be conducted.
Sponsor: Boston Medical Center (Other)
Collaborators: Wagner Foundation (Unknown); Someone Elses Child (Unknown); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-43633
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Financial Hardship; Food Insecurity; Health Status
Keywords: Financial insecurity; Food insecurity; Health Status; Mental Health Assessment; Mental Health
MeSH Terms: conditions — Financial Stress; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Step wedge design: participants randomized in two groups, Group 1, and Group 2 - intervention on different timeframe, analysis of the difference and similarities between groups pre- and post-survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Career Navigator Coaching (Other): Participants randomized into this group will be invited to participate in the quantitative and qualitative surveys. At baseline, participants in Group1 will receive the intervention- tailored coaching sessions with the Career Navigator which will continue until the end of the 6th month.
  The intervention will be tailored for each participant according to their need. The Career Navigator will be in charge to plan and develop tools to help the participant achieve their own goals.
  Interventions: Behavioral: Career Navigator Coaching
- Delayed Career Navigator Coaching (Other): Participants randomized into this group will be invited to participate in the quantitative and qualitative surveys For the first six months, participants in Groups 2 will not receive the intervention and will function as a control group. When the study reaches the sixth-month Group 2 participants will receive the intervention - tailored coaching sessions with the Career Navigator.
  The intervention will be tailored for each participant according to their need. The Career Navigator will be in charge to plan and develop tools to help the participant achieve their own goals.
  Interventions: Behavioral: Career Navigator Coaching

INTERVENTIONS:
Behavioral: Career Navigator Coaching — The Career Navigator will support participants with a tailored approach to reach career and financial goals through one or more of the following services, in addition to referrals to other external services (community-based organizations) as needed for 6 months:
  1. Career pathway navigation
  2. Employee benefit maximization
  3. Financial literacy and wealth building
  4. Services funds for resources that mitigate specific barriers or needs.

SUMMARY:
Research on economic mobility barriers consistently demonstrates that lack of access to jobs that pay living wages and to asset building opportunities coupled with cliff effects across public assistance programs (families losing multiple benefits at the same time when their incomes increase) traps families in a cycle of poverty and food insecurity, and as a result, negatively impacts their financial well-being and physical and mental health.

The investigators will explore the extent to which an Economic Mobility Pilot improves the financial well-being, physical and mental health, and reduces the social risks of study participants. Study participants will be eligible consented Boston Medical Center (BMC) employees.

The intervention developed for this study consists of six months of coaching session offered by the Career Navigator. Participant will receive support on career and financial through services, such as career pathway navigation, employee benefit maximization, financial literacy, wealth building, resources, and referrals.

A step wedge design will be implemented with participants randomized in two groups, Group 1, and Group 2 - intervention on different timeframe, analysis of the difference and similarities between groups pre- and post-survey. The qualitative component will include focus group of participants to provide information on the employee's perception of the intervention received, barriers to adherence and facilitators, and semi- structured interviews of the employer leadership to help assess the barriers and facilitators of the pilot.

A primary aim of this research is to monitor changes in economic mobility and financial well-being. Additional aims are to investigate changes in household hardships and employee, employee depressive symptoms, and their child's health. The investigators will examine whether the participants in the intervention group compared to those before receiving the intervention, are more likely to:

* Increase employee retention and self-reported financial well-being.
* Improve self-reported food security.
* Improve housing stability, energy security, childcare access, and/or health care access.
* Improve employee self-reported physical health status, and/or reduce self-reported anxiety and depressive symptoms.
* Improve employee-reported physical health status of the employee's child.
* Cost of delivery of the intervention
* Increased family income as result of this intervention

DETAILED DESCRIPTION:
During the COVID-19 pandemic longstanding economic inequities have been exacerbated for people with low incomes in frontline and service sector jobs. These inequities are manifested downstream in the form of food insecurity (FI) and related health consequences. Research on economic mobility barriers consistently demonstrates that lack of access to jobs that pay living wages and to asset building opportunities coupled with cliff effects across public assistance programs (families losing multiple benefits at the same time when their incomes increase) traps families in a cycle of poverty and economic hardships, and as a result, negatively impacts their physical and mental health. This study proposes to explore the extent to which an Economic Mobility Pilot improves the financial well-being, physical and mental health, and reduces the social risks of study participants.

As part of Boston Medical Center (BMC) commitment to advancing its mission to promote equity as an anchor institution in the community, the health system seeks to identify strategies that increase employment and career building opportunities for members of marginalized communities served by BMC. The Boston Collaborative plays a leading role in advancing these goals and has deeply engaged community-led organizations and members, as well as local and hospital leadership to identify economic mobility pathways and place-based solutions that are responsive to the needs of specific communities.

Social capital, the connections to people and information, increases individuals' overall well-being and ability to both give and receive a range of supports that promote positive outcomes for caregivers and their children. By providing social capital, financial resources, and benefit maximization, this pilot will maximize assistance benefit; improve financial well-being and job retention. The participants may receive additional services, which could increase quality of life.

Social capital will be increased in participants through the intervention which is six months of tailored coaching session offered by the Career Navigator. The Career Navigator will meet (either in person or online) with the participant and offer support with career planning and development, employee benefit maximization, financial well-being and management, flex fund access, and other resources.

The quantitative component of this pilot will help the investigators better understand barriers and facilitators of economic mobility from the employee and employer perspectives. The participant employees will help with lessons learned through the development and implementation of the pilot, participant adherence, and challenges. The participant employer leaders will help with best practices, challenges, adaptation, and innovations.

About 60 Boston Medical Center (BMC) employees living in one of the following seven zip codes (02119, 02121, 02122, 02124, 02125, 02126, 02130) will be invited to participate in this study.

Survey instruments consist of valid and reliable scales which will be used to collect information on demographics, financial well-being, economic mobility, food security, housing security, health care utilization, child health outcomes, child development, employee physical and mental health. See attached survey instrument for detailed research questions.

Surveys conducted after baseline will consist of questions regarding social determinants of health, financial well-being, and economic mobility. Will not include variables, such as demographics, that would remain unchanged from one time to the next.

The baseline survey contains questions related to demographics, food security, housing stability, and participant physical and mental health, child health, childcare, participation in programs, financial well-being, and economic mobility.

Between data collection periods, (baseline, 3, 6, 9, 12 and 18 months of enrollment), subjects will be working with the Career Navigator, who will build with each participant tools and resources customized to their needs. The intervention with the Career Navigator will have a total duration of 6 months for each of the study arms (Group 1 and Group 2).

Baseline, the 6-month, 12-month and the 18-month, all individuals will be approached to participate in a survey. At Baseline, the Group 1 starts the intervention. At the 6-month, Group 1 finalizes intervention meanwhile Group 2 starts intervention, which finalizes at 12-month. At the 3- and the 9-month, all participants will be approached for qualitative focus groups and a quarterly check-in. At the 18-month, all the individuals will be approached for the final survey.

ELIGIBILITY:
Newly hired Boston Medical Center (hires since 2021) employees with children from the seven historically marginalized zip codes in Boston (mainly in the neighborhoods of Roxbury, Dorchester, and Mattapan) receiving hourly rate less than $35.00.

Inclusion Criteria:

* Recently hired Boston Medical Center employees, since June 2021
* Employees financially responsible for a child 18 years of age or younger
* Employees who live in one of the following zip codes: 02119, 02121, 02122, 02124, 02125, 02126, 02130
* Employees who have Income threshold hourly wage of $35 Dollars

Exclusion Criteria:

* Employees who have been previously contacted by the Career Navigator
* Employees not financially responsible for a child of 18 years old of age or younger
* Employees not interested in receiving support from Career Navigator
* Employees who do not accept consent
* Employees who Do not reside in one of the seven zip codes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Financial well-being | 18 months
  Financial well-being will be assessed using the Consumer Financial Protection Bureau's abbreviated 5-item scale, covering aspects such as income, employment, savings, safety net, past financial experiences, and financial behaviors, skills, and attitudes. Ratings will be given on a scale from 0 to 4, indicating the level of description or frequency, with higher values representing stronger agreement or more frequent occurrences. The collected scores will be aggregated and categorized by age and administration type (self or external). The Item Response Theory (IRT) model will be employed to ensure the validity and significance of the items, while a higher score on the scale will reflect greater financial security.
Food insecurity | 18 months
  Food security status over the past year will be assessed using the validated Abbreviated Child and Adult Food Security Scale (ACAFSS), which includes 6 household-specific and 2 child-specific questions. Household are classified into 3 categories: (1) household food secure (HFS) if one or none questions were endorsed as sometimes or often true, (2) household FI (HFI) if three or more, or the 4th question on household were endorsed, and (3) child FI if 2 or more child-specific questions were endorsed.

SECONDARY OUTCOMES:
Housing instability | 18 months
  Participants will be categorized as experiencing housing insecurity (HI) if they report (1) being behind on rent/mortgage in the past year, (2) moving 2 or more times in the past year, and/or (3) homelessness within the child's lifetime.
Child Health Outcomes | 18 months
  Child health status will be characterized by caregiver rating of child health as excellent, good, fair, or poor, using a question from the National Health and Nutrition Examination Survey (NHANES).
Lifetime Child Hospitalizations | 18 months
  This outcome will be assessed by a question asked to the caregiver. Any hospitalizations will be defined as ≥1 hospitalizations in the child's lifetime, excluding the birth hospitalization.
Participant Health Outcomes | 18 months
  Child and subject general health status will be reported by the participating using validated questions from National Health and Nutrition Examination Survey (NHANES).
Parental depressive symptoms | 18 months
  Parental depressive symptoms will be collected using the Patient Health Questionnaire-2 (PHQ-2) which is a 2 question instrument with potential responses from 0 to 3 where 0=Not at all, 1=Several days, 2= More than half the days, and 4=Nearly every day. PHQ-2 scores range from 0-6. If the score is 3 or greater, major depressive disorder is likely.
Public program participation | 18 months
  Participants will be asked "yes or no" question on the following programs participation: Woman Infant and Child Program (WIC), Supplemental Nutrition Assistance Program (SNAP), and Transitional Aid to Families Needy Families (TANF). Medicaid, Earned Income Tax Credit (EITC), Subsidized housing or public housing, Energy Assistance, Water Assistance, Social Security (SSI) Disability Benefits (SSDI), Head Start or Early Start services, Free or reduced priced schools meals, Summer Meals, Childcare subsidy or voucher, Unemployment insurance, Electronic Benefit Transfer (EBT).

CONTACTS AND LOCATIONS:
Overall Officials: Megan Sandel, MD MPH, Principal Investigator — Boston Medical Center and Boston University Chobanian
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Bethell CD, Read D, Stein RE, Blumberg SJ, Wells N, Newacheck PW. Identifying children with special health care needs: development and evaluation of a short screening instrument. Ambul Pediatr. 2002 Jan-Feb;2(1):38-48. doi: 10.1367/1539-4409(2002)0022.0.co;2. PMID 11888437
- [Background] Woolfenden S, Eapen V, Williams K, Hayen A, Spencer N, Kemp L. A systematic review of the prevalence of parental concerns measured by the Parents' Evaluation of Developmental Status (PEDS) indicating developmental risk. BMC Pediatr. 2014 Sep 13;14:231. doi: 10.1186/1471-2431-14-231. PMID 25218133
- [Background] Sandel M, Sheward R, Ettinger de Cuba S, Coleman SM, Frank DA, Chilton M, Black M, Heeren T, Pasquariello J, Casey P, Ochoa E, Cutts D. Unstable Housing and Caregiver and Child Health in Renter Families. Pediatrics. 2018 Feb;141(2):e20172199. doi: 10.1542/peds.2017-2199. Epub 2018 Jan 22. PMID 29358482
- [Background] Kemper KJ, Babonis TR. Screening for maternal depression in pediatric clinics. Am J Dis Child. 1992 Jul;146(7):876-8. doi: 10.1001/archpedi.1992.02160190108031. PMID 1496962
- [Background] Glascoe FP. Evidence-based approach to developmental and behavioural surveillance using parents' concerns. Child Care Health Dev. 2000 Mar;26(2):137-49. doi: 10.1046/j.1365-2214.2000.00173.x. PMID 10759753
- [Background] Ettinger de Cuba S, Chilton M, Bovell-Ammon A, Knowles M, Coleman SM, Black MM, Cook JT, Cutts DB, Casey PH, Heeren TC, Frank DA. Loss Of SNAP Is Associated With Food Insecurity And Poor Health In Working Families With Young Children. Health Aff (Millwood). 2019 May;38(5):765-773. doi: 10.1377/hlthaff.2018.05265. PMID 31059367
- [Background] Cook JT, Frank DA, Casey PH, Rose-Jacobs R, Black MM, Chilton M, Ettinger de Cuba S, Appugliese D, Coleman S, Heeren T, Berkowitz C, Cutts DB. A brief indicator of household energy security: associations with food security, child health, and child development in US infants and toddlers. Pediatrics. 2008 Oct;122(4):e867-75. doi: 10.1542/peds.2008-0286. PMID 18829785
- [Background] O'Hara B, Caswell K. Health Status, Health Insurance, and Medical Services Utilization: 2010. Household Economic Studies. Washington, DC: US Census Bureau. 2013.
- [Background] Falci SG, Marques LS. CONSORT: when and how to use it. Dental Press J Orthod. 2015 May-Jun;20(3):13-5. doi: 10.1590/2176-9451.20.3.013-015.ebo. No abstract available. PMID 26154451
- [Background] Bailey MJ, DiNardo J, Stuart BA. THE ECONOMIC IMPACT OF A HIGH NATIONAL MINIMUM WAGE: EVIDENCE FROM THE 1966 FAIR LABOR STANDARDS ACT. J Labor Econ. 2021 Apr;39(Suppl 2):S329-S367. doi: 10.1086/712554. PMID 35414741